CLINICAL TRIAL: NCT00972504
Title: A Randomised, Double-blind, Placebo-controlled 4-period Cross-over Study to Assess the Efficacy and Safety of Repeat Dose Intranasal GSK1004723 (1000µg), Oral GSK835726 (10mg) and Cetirizine (10mg) in the Environmental Challenge Chamber in Subjects With Seasonal Allergic Rhinitis
Brief Title: 723/726 Proof of Concept Study in Allergen Challenge Chamber in Hannover
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 112864
Record Dates: First submitted 2009-08-27; First posted 2009-09-07 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-03

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Proof of concept
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — GSK 835726; GSK 1004723; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK835726 (10mg) (Active Comparator): 10mg oral dose
  Interventions: Drug: GSK835726 10mg
- GSK1004723 (1000mcg) (Active Comparator): 1000mcg nasal spray solution
  Interventions: Drug: GSK1004723 1000mcg
- Cetirizine 10mg (Active Comparator): 10mg cetirizine as active comparator
  Interventions: Drug: Cetirizine 10mg
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GSK835726 10mg — GSK835726 10mg tablet
  Arms: GSK835726 (10mg)
Drug: GSK1004723 1000mcg — GSK1004723 1000mcg nasal spray solution
  Arms: GSK1004723 (1000mcg)
Drug: Cetirizine 10mg — Cetirizine 10mg active comparator
  Arms: Cetirizine 10mg
Drug: placebo — placebo to match actives
  Arms: placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled 4-period cross-over study to assess the efficacy and safety of repeat dose intranasal GSK1004723 (1000µg), oral GSK835726 (10mg) and cetirizine (10mg) in the environmental challenge chamber in subjects with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy apart from seasonal allergic rhinitis, as determined by a physician. Can have mild asthma.
* Males or female using contraceptives
* Aged 18 - 65
* Weight 50kg+, BMI 19-32 kg/m2
* Exhibit response to Challenge Chamber and skin prick test.
* Non-smoker
* Capable of giving informed consent
* AST and ALT<2xULN; alkaline phosphatase and bilirubin <or=1.5xULN

Exclusion Criteria:

* No nasal structural abnornmality/polyposis, surgery, infection.
* any respiratory disease, other than mild asthma or seasonal allergic rhinitis
* participated in another clinical study within 30 days.
* Subject has donated a unit of blood within 1 month
* Use of prescription or non-prescription drugs, including vitamins and st john's wort within 7 days of trial.
* History of sensitivty to drug
* History of alcohol/drug abuse within 12 months.
* Positive Hepatitis B antibody test
* Positive HIV antibody test
* Risk of non-compliance with study protocol
* Pregnant or llactating females
* Perenial allergic rhinitis
* Administration of oral, injectable or dermal corticosteriods within 8 weeks, intranasal or inhaled within 3 weeks.
* Past or present disease that may affect outcome, as judge by investigator
* Specific Immunotherapy within 2 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-06-01; Primary Completion 2009-08-01 (Actual); Study Completion 2009-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Daley-Yates P, Ambery C, Sweeney L, Watson J, Oliver A, McQuade B. The efficacy and tolerability of two novel H(1)/H(3) receptor antagonists in seasonal allergic rhinitis. Int Arch Allergy Immunol. 2012;158(1):84-98. doi: 10.1159/000329738. Epub 2011 Dec 29. PMID 22212854
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 112864 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112864 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112864 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112864 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112864 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112864 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112864 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June-2009 to August-2009, total of 54 participants were randomized at one site in Germany.
Pre-assignment Details: All participants had a diagnosis of seasonal allergic rhinitis and exhibited a moderate response to allergen challenge in the environmental challenge chamber (ECC) at Screening, defined as total nasal symptom score (TNSS) more than equal to (>=) 6.
Groups:
- Overall Study: Participants randomized to receive once daily GSK1004723 (1000 micrograms [µg]) nasal spray solution for 3 days or oral tablet of GSK835726 (10 milligram [mg]) or oral capsule of cetirizine (10 mg) or matching placebo of these investigational products as per randomization schedule in the morning of each day. Each participant dosed at the same time each day relative to Day 1. Each treatment period was separated by at least 4 days washout period and there was at least 7 days between ECC days.
Period: Overall Study
Arm/Group | Overall Study
Started | 54
Completed | 51
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Investigator discretion | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Participants randomized to receive once daily GSK1004723 1000 µg nasal spray solution for 3 days or oral tablet of GSK835726 10 mg or oral capsule of cetirizine 10 mg or matching placebo of these investigational products as per randomization schedule in the morning of each day. Each participant dosed at the same time each day relative to Day 1. Each treatment period was separated by at least 4 days washout period and there was at least 7 days between ECC days.
Arm/Group | Overall Study
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 39
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 54

OUTCOME MEASURES:

1. Primary Outcome: Weighted Mean TNSS (Sneeze, Itch, Rhinorrhoea and Nasal Blockage) 1-6 Hours Post Start of Allergen Challenge (2-7 Hours Post-dose) on Day 3
Description: On the third dosing day, participants entered the ECC for a duration of 6 hours, 1 hour after receiving their third dose. Time 0 hour was considered as the time that the participant entered the ECC. Nasal blockage, itch, sneeze and rhinorrhoea was scored on a categorical scale from 0 to 3 (0: no symptoms; 1: mild symptoms; 2: moderate symptoms; 3: severe symptoms). The total TNSS ranged from 0-12 point, with low score indicates well-being and higher score indicates more severity. Individual symptoms scores was summed at each time point (0, 20, 40, 60, 80, 100, 120, 140, 160, 180, 200, 220, 240, 260, 280, 300, 320, 340 and 360 minutes). The adjusted mean is provided as least square mean.
Time Frame: Day 3 of each treatment period (approximately up to 63 days)
Population: The all subjects population was used defined as all participants who receive at least one dose of study medication. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Placebo: Participants randomized to this arm received placebo once daily for 3 days (to match GSK1004723, GSK835726 and cetirizine) as per randomization schedule in the morning of each day. Each participant dosed at the same time each day relative to Day 1. Each treatment period was separated by at least 4 days washout period and there was at least 7 days between ECC days.
- GSK1004723 1000 µg Once Daily: Participants randomized to this arm received once daily GSK1004723 1000 µg nasal spray solution for 3 days, plus placebos to match both GSK835726 and cetirizine as per randomization schedule in the morning of each day. Each participant dosed at the same time each day relative to Day 1. Each treatment period was separated by at least 4 days washout period and there was at least 7 days between ECC days.
- GSK835726 10 mg Once Daily: Participants randomized to this arm received once daily oral tablet of GSK835726 10 mg for 3 days, plus placebos to match both GSK1004723 and cetirizine as per randomization schedule in the morning of each day. Each participant dosed at the same time each day relative to Day 1. Each treatment period was separated by at least 4 days washout period and there was at least 7 days between ECC days.
- Cetirizine 10 mg Once Daily: Participants randomized to this arm received once daily oral capsule of cetirizine 10 mg for 3 days, plus placebos to match both GSK1004723 and GSK835726 as per randomization schedule in the morning of each day. Each participant dosed at the same time each day relative to Day 1. Each treatment period was separated by at least 4 days washout period and there was at least 7 days between ECC days.
Arm/Group | Placebo | GSK1004723 1000 µg Once Daily | GSK835726 10 mg Once Daily | Cetirizine 10 mg Once Daily
Number analyzed (Participants) | 51 | 53 | 53 | 51
Score on a scale | 4.9 [4.4 to 5.4] | 4.2 [3.7 to 4.8] | 3.6 [3.1 to 4.1] | 3.5 [3.0 to 4.1]
Statistical Analysis 1: Comparison: Placebo vs GSK1004723 1000 µg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.2 to -0.1], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs GSK835726 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-1.8 to -0.8], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Placebo vs Cetirizine 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-1.9 to -0.8], Standard Error of Mean 0.27

2. Secondary Outcome: Weighted Mean of the Individual Components of TNSS (Sneeze, Itch, Rhinorrhoea and Nasal Blockage) 1-6 Hours Post Start of Allergen Challenge (2-7 Hours Post-dose) on Day 3
Description: On the third dosing day, participants entered the ECC for a duration of 6 hours, 1 hour after receiving their third dose. Time 0 hour was considered as the time that the participant entered the ECC. Nasal blockage, itch, sneeze and rhinorrhoea was scored on a categorical scale from 0 to 3 (0: no symptoms; 1: mild symptoms; 2: moderate symptoms; 3: severe symptoms). The total TNSS ranged from 0-12 point, with low score indicates well-being and higher score indicates more severity. Individual symptoms scores was summed to produce the TNSS at each time point (0, 20, 40, 60, 80, 100, 120, 140, 160, 180, 200, 220, 240, 260, 280, 300, 320, 340 and 360 minutes). The adjusted mean is provided as least square mean.
Time Frame: Day 3 of each treatment period (approximately up to 63 days)
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | GSK1004723 1000 µg Once Daily | GSK835726 10 mg Once Daily | Cetirizine 10 mg Once Daily
Number analyzed (Participants) | 51 | 53 | 53 | 51
Score on a scale
  Nasal Blockage | 1.5 [1.3 to 1.7] | 1.7 [1.5 to 1.8] | 1.3 [1.1 to 1.4] | 1.3 [1.1 to 1.4]
  Rhinorrhoea | 1.5 [1.3 to 1.7] | 1.3 [1.1 to 1.4] | 1.1 [0.9 to 1.3] | 1.0 [0.9 to 1.2]
  Nasal Itching | 1.1 [0.9 to 1.3] | 0.9 [0.7 to 1.0] | 0.8 [0.6 to 1.0] | 0.8 [0.6 to 1.0]
  Sneezing | 0.8 [0.7 to 0.9] | 0.4 [0.3 to 0.6] | 0.5 [0.4 to 0.6] | 0.5 [0.3 to 0.6]
Statistical Analysis 1: Comparison: Placebo vs GSK1004723 1000 µg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.0 to 0.3], Standard Error of Mean 0.09 — Comparison of Nasal Blockage between Placebo and GSK1004723 1000 µg once daily
Statistical Analysis 2: Comparison: Placebo vs GSK835726 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.09 — Comparison of Nasal Blockage between Placebo and GSK835726 10 mg once daily
Statistical Analysis 3: Comparison: Placebo vs Cetirizine 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.09 — Comparison of Nasal Blockage between Placebo and Cetirizine 10 mg once daily
Statistical Analysis 4: Comparison: Placebo vs GSK1004723 1000 µg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.08 — Comparison of Rhinorrhoea between Placebo and GSK1004723 1000 µg once daily
Statistical Analysis 5: Comparison: Placebo vs GSK835726 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2], Standard Error of Mean 0.08 — Comparison of Rhinorrhoea between Placebo and GSK835726 10 mg once daily
Statistical Analysis 6: Comparison: Placebo vs Cetirizine 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.6 to -0.3], Standard Error of Mean 0.08 — Comparison of Rhinorrhoea between Placebo and Cetirizine 10 mg once daily
Statistical Analysis 7: Comparison: Placebo vs GSK1004723 1000 µg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.08 — Comparison of Nasal Itching between Placebo and GSK1004723 1000 µg once daily
Statistical Analysis 8: Comparison: Placebo vs GSK835726 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.2], Standard Error of Mean 0.08 — Comparison of Nasal Itching between Placebo and GSK835726 10 mg once daily
Statistical Analysis 9: Comparison: Placebo vs Cetirizine 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.2], Standard Error of Mean 0.08 — Comparison of Nasal Itching between Placebo and Cetirizine 10 mg once daily
Statistical Analysis 10: Comparison: Placebo vs GSK1004723 1000 µg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.2], Standard Error of Mean 0.07 — Comparison of Sneezing between Placebo and GSK1004723 1000 µg once daily
Statistical Analysis 11: Comparison: Placebo vs GSK835726 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.4 to -0.2], Standard Error of Mean 0.07 — Comparison of Sneezing between Placebo and GSK835726 10mg once daily
Statistical Analysis 12: Comparison: Placebo vs Cetirizine 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.2], Standard Error of Mean 0.07 — Comparison of Sneezing between Placebo and Cetirizine 10mg once daily

3. Secondary Outcome: Weighted Mean Wet Tissue Weight (as a Surrogate Marker of Nasal Secretion) 1-6 Hours Post Start of Allergen Challenge (2-7 Hours Post-dose) on Day 3
Description: On the third dosing day, participants entered the ECC for a duration of 6 hours, 1 hour after receiving their third dose. Time 0 hour was considered as the time that the participant entered the ECC. Wet tissue weight assessments was measured as a surrogate marker of nasal secretion at 60, 120, 180, 240, 300 and 360 minutes. The adjusted mean is provided as least square mean.
Time Frame: Day 3 of each treatment period (approximately up to 63 days)
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Grams
Arm/Group | Placebo | GSK1004723 1000 µg Once Daily | GSK835726 10 mg Once Daily | Cetirizine 10 mg Once Daily
Number analyzed (Participants) | 51 | 53 | 53 | 51
Grams | 6.251 [5.198 to 7.304] | 5.210 [4.167 to 6.254] | 4.491 [3.446 to 5.536] | 3.459 [2.406 to 4.512]
Statistical Analysis 1: Comparison: Placebo vs GSK1004723 1000 µg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -1.041, 95% CI 2-sided [-1.870 to -0.212], Standard Error of Mean 0.4194
Statistical Analysis 2: Comparison: Placebo vs GSK835726 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -1.760, 95% CI 2-sided [-2.584 to -0.936], Standard Error of Mean 0.4172
Statistical Analysis 3: Comparison: Placebo vs Cetirizine 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -2.792, 95% CI 2-sided [-3.626 to -1.957], Standard Error of Mean 0.4224

4. Secondary Outcome: Weighted Mean Nasal Congestion VAS 1-6 Hours Post Start of Allergen Challenge (2-7 Hours Post-dose) on Day 3
Description: On the third dosing day, participants entered the ECC for a duration of 6 hours, 1 hour after receiving their third dose. Time 0 hour was considered as the time that the participant entered the ECC. Nasal congestion was measured on 0-10 centimeter VAS scale (0: no symptoms and 10: the worst possible symptoms) with low score indicates well-being and higher values indicate greater congestion. It was measured at 60, 80, 100, 120, 140, 160, 180, 200, 220, 240, 260, 280, 300, 320, 340 and 360 minutes. The adjusted mean is provided as least square mean.
Time Frame: Day 3 of each treatment period (approximately up to 63 days)
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | GSK1004723 1000 µg Once Daily | GSK835726 10 mg Once Daily | Cetirizine 10 mg Once Daily
Number analyzed (Participants) | 51 | 53 | 53 | 51
Score on a scale | 3.97 [3.36 to 4.57] | 4.29 [3.69 to 4.89] | 2.92 [2.32 to 3.52] | 2.90 [2.29 to 3.51]
Statistical Analysis 1: Comparison: Placebo vs GSK1004723 1000 µg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.28 to 0.93], Standard Error of Mean 0.306
Statistical Analysis 2: Comparison: Placebo vs GSK835726 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.65 to -0.45], Standard Error of Mean 0.305
Statistical Analysis 3: Comparison: Placebo vs Cetirizine 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Final Values) = -1.07, 95% CI [-1.68 to -0.46], Standard Error of Mean 0.308

5. Secondary Outcome: Mean Forced Expiratory Volume in 1 Second (FEV1)
Description: On the third dosing day, participants entered the ECC for a duration of 6 hours, 1 hour after receiving their third dose. Time 0 hour was considered as the time that the participant entered the ECC. FEV1 was measured at pre-challenge, 60, 120, 180, 240, 300 and 360 minutes.
Time Frame: Day 3 of each treatment period (approximately up to 63 days)
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed (represented by n=x,x,x,x,x in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the All Subjects population.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | GSK1004723 1000 µg Once Daily | GSK835726 10 mg Once Daily | Cetirizine 10 mg Once Daily
Number analyzed (Participants) | 52 | 54 | 53 | 52
Liters
  FEV1-Pre challenge: number analyzed (Participants) | 51 | 53 | 53 | 52
  FEV1-Pre challenge | 3.908 (0.7051) | 3.935 (0.6515) | 3.924 (0.7055) | 3.932 (0.6654)
  FEV1,1 hour: number analyzed (Participants) | 51 | 53 | 53 | 52
  FEV1,1 hour | 3.949 (0.7319) | 3.959 (0.6804) | 3.948 (0.7125) | 3.958 (0.6865)
  FEV1,2 hour: number analyzed (Participants) | 51 | 53 | 53 | 51
  FEV1,2 hour | 3.910 (0.7161) | 3.948 (0.6444) | 3.936 (0.7014) | 3.925 (0.6829)
  FEV1,3 hour: number analyzed (Participants) | 51 | 53 | 53 | 51
  FEV1,3 hour | 3.901 (0.7134) | 3.938 (0.6774) | 3.918 (0.6941) | 3.899 (0.7179)
  FEV1,4 hour: number analyzed (Participants) | 51 | 53 | 53 | 51
  FEV1,4 hour | 3.881 (0.7364) | 3.913 (0.7083) | 3.903 (0.7067) | 3.903 (0.7124)
  FEV1,5 hour: number analyzed (Participants) | 51 | 53 | 53 | 51
  FEV1,5 hour | 3.858 (0.7314) | 3.890 (0.6868) | 3.890 (0.6954) | 3.858 (0.7406)
  FEV1,6 hour: number analyzed (Participants) | 50 | 53 | 53 | 51
  FEV1,6 hour | 3.914 (0.7099) | 3.877 (0.6381) | 3.887 (0.6894) | 3.868 (0.7231)

6. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or is associated with liver injury and impaired liver function defined as: alanine aminotransferase >=3 times upper limit of normal (ULN), and total bilirubin >=2 times ULN or international normalized ratio more than 1.5.
Time Frame: approximately up to 63 days
Population: All Subjects population.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK1004723 1000 µg Once Daily | GSK835726 10 mg Once Daily | Cetirizine 10 mg Once Daily
Number analyzed (Participants) | 52 | 54 | 53 | 52
Participants
  Any AE | 15 | 53 | 13 | 17
  Any SAE | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were reported throughout the study (approximately up to 63 days).
Description: All subject population was used.
Arm/Group | Placebo | GSK1004723 1000 µg Once Daily | GSK835726 10 mg Once Daily | Cetirizine 10 mg Once Daily
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/54 | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/54 | 0/53 | 0/52
Other Adverse Events (participants affected / at risk) | 15/52 | 53/54 | 13/53 | 17/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | GSK1004723 1000 µg Once Daily (N=54) | GSK835726 10 mg Once Daily (N=53) | Cetirizine 10 mg Once Daily (N=52)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 47 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 8 | 7 | 6 | 11
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Hypotonia (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 4 | 3 | 4
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 5 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Forced expiratory volume decreased (Investigations) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.